CLINICAL TRIAL: NCT05109143
Title: Efficacy of Rectal Indomethacin in Prevention of Post-operative Pancreatitis After Pancreaticoduodenectomy - a Randomized Controlled Trial
Brief Title: Efficacy of Rectal Indomethacin in Prevention of Post-operative Pancreatitis After Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEC/2020/81/MA13
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-10

CONDITIONS: Pancreatoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B (Active Comparator): Standard Medical Treatment
  Interventions: Other: Standard Medical Treatment
- Group A (Experimental): Will be administered 100mg of Indomethacin Suppository sigle dose at the time of induction of anesthesia with Standard Medical Treatment
  Interventions: Drug: Indomethacin suppository; Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Indomethacin suppository — 100mg Indomethacin Suppository administered at the time of Induction
  Arms: Group A
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Pancreatico-duodenectomy is one of the commonly performed procedure for periampullary/distal cholangio/head of pancreas carcinoma. Post operative pancreatitis is an emerging concept, recently being studied as one of the most important contributing factor of Post-operative pancreatic fistula, which is one of the major complication of pancreatoduodenectomy. Rectal indomethacin, a type of non-steroidal anti-inflammatory drug, when given in a single dose has been shown to prevent pancreatitis in patients undergoing ERCP. In this study, we will be administering rectal indomethacin at the time of induction of anesthesia to the experimental arm of the study and compare the results in terms of incidence of post-operative pancreatitis in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All consenting adults planned to undergo pancreatoduodenectomy,

Exclusion Criteria:

* asthma
* allergic reactions to NSAIDs
* CKD
* internal hemorrhoids
* anti-platelet medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Post-operative Pancreatitis | first 30 days following pancreatoduodenectomy

SECONDARY OUTCOMES:
Post-operative Pancreatic Fistula | first 30 days following pancreatoduodenectomy
delayed gastric emptying | First 30 days following pancreatoduodenectomy
intra-abdominal abscess | first 30 days following pancreatoduodenectomy
Length of ICU stay | First 30 days following pancreatoduodenectomy
Length of hospital stay | First 30 days following pancretoduodenectomy
risk factors of post-operative pancreatitis | first 30 days following pancreatoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, FEBS, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No